CLINICAL TRIAL: NCT03651570
Title: Implementing an e-Intervention to Reduce Anxiety Symptoms and Improve Psychosocial Oncology Uptake in Patients Newly Diagnosed With Head and Neck Cancer: Pilot Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of a E-intervention to Help Patients Newly Diagnosed With Cancer Cope Better: Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Melissa Henry, Principal Investigator, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MM-CODIM-FLP-17-085
Record Dates: First submitted 2018-06-26; First posted 2018-08-29 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PTSD Coach (Experimental): PTSD Coach is a mobile mental health app developed by US Veterans Affairs translated into French by Veterans Affairs Canada in partnership with the Department of National Defence and the Canadian Mental Health Association. It was developed for a male population (92% of veterans are men), as is predominantly found in HNC, and addresses the issue of mental health and stigma as found in our HNC patients. PTSD Coach can be used as a stand-alone education and symptom management and contains 4 modules: 1) Learn- Module, 2) Self-Assessment-Module, 3) Manage Symptoms-Module and 4) Find Support-Module. The content of the first and last modules were adapted to the oncological population.
  Interventions: Device: PTSD Coach
- Game application (Placebo Comparator): Patients will be assigned to three apps involving playing a game (i.e., Candy Crush, Tetris, or Solitaire), during the waiting time before and between medical treatments in the hospital, on the same weekly schedule as the experimental group. The game apps contain no element of intervention and were selected based on popularity and capacity to interests.
  Interventions: Behavioral: Game application
- Usually Care Control Group (No Intervention): The Otolaryngology - Head and Neck Surgery (OHNS) Departments do not offer systematic interventions on anxiety and self-management, neither does any intervention address stigma. However, participating recruitment centres are already offering a best-of-care approach with well-established psychosocial oncology services, including psychiatrists, psychologists, social workers, nurses, and volunteers. All participants will be free to use hospital- or community-based support throughout the study, which will be tracked in all groups via questionnaire and chart review.

INTERVENTIONS:
Device: PTSD Coach — PTSD Coach is a mobile mental health app that addresses the issue of mental health and stigma which can be used as a stand-alone education and symptom management and contains 4 modules: 1) Learn- Module, 2) Self- Assessment-Module, 3) Manage Symptoms-Module and 4) Find Support-Module.
  Arms: PTSD Coach
Behavioral: Game application — This control condition is important to control for distraction (attention on something pleasant or a task) and the human factor involved in usage prompting (i.e., same exposure time + contacts with personnel), since either distraction or the human contact with staff may, alone, lower anxiety
  Arms: Game application

SUMMARY:
Informed by a previous trial in general cancer patients, the investigators aim to conduct a multi-centre Phase III explanatory RCT to demonstrate a significant impact of PTSD Coach on levels of anxiety in head and neck cancer (HNC) patients, including saliva and hair cortisol as bio-immunological indicators for stress. However, prior to proposing a larger trial requiring 267 patients, the investigators aim to demonstrate feasibility of recruitment and compliance with protocol procedures in a Phase II Pilot of 60 newly diagnosed HNC patients. The EG will receive PTSD Coach + usual care, compared to two control groups (UC and AC). AC will be comprised of a game app (e.g., Tetris, Candy Crush, or Solitaire) and will be structurally equivalent to the EG to control for distraction (attention on something pleasant or a task) and the human factor involved in usage prompting (i.e., same exposure time + contacts with personnel), since either distraction or the human contact with staff may, alone, lower anxiety. From a resource allocation perspective, it is important to know if the positive effects of PTSD Coach are due to the intervention itself or to the use of an app and its usage prompting. The investigators believe that PTSD Coach will be even more effective at reducing anxiety in HNC patients, as it teaches specific CBT techniques and uses psychoeducation already found to be more effective than distraction alone.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with HNC (all HNC sites; TNM classification system); first occurrence, progression or recurrence <4 weeks at referral.
2. Willing to complete PTSD Coach or game app within 3 weeks as they await treatment onset.
3. >18 years old
4. Alert and capable of giving free and informed consent according to referring clinician.

Exclusion Criteria:

1. Karnofsky Performance Status (KPS) score < 60 (rated by referring oncologists/nurses or Research Coordinator) or expected survival <6 months according to clinical judgment of physicians and/or nurses.
2. Suicidal. Present a score of ≥2 on the Beck Depression Inventory (BDI) suicide item.
3. Known diagnosis of schizophrenia or schizoaffective disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment for a full trial study | 2 months post-randomization
  1. Can we recruit a sufficient number (i.e., n=60 over 8 months or 8/month) of newly diagnosed head and neck cancer patients? AND
  2. Can we retain a sufficient proportion (i.e., ≥85% at three months post-randomization, having completed the primary outcome) of head and neck patients in all trial arms to allow completion of a full study (n=267) in a timely fashion?
PTSD Coach app Acceptability | 2 months post-randomization
  Is the PTSD Coach app acceptable to at least 80% of newly diagnosed head and neck cancer patients, as indicated by 80% positive responses on the Pilot-Study Questionnaire (PSQ; adapted from the CSQ-8; Attkisson & Zwick, 1982)

SECONDARY OUTCOMES:
Completion of intervention in a timely manner | 2 months post-randomization
  At least 90% of experimental group complete PTSD Coach within 3 weeks from randomization.
  At least 85% of the content for each module of PTSD Coach be completed.
  At least 90% of the attention control complete their assigned condition as planned (i.e., 45 min/week over 3 weeks).
Sample size calculation for full trial study | 2 months post-randomization
  Identify the 80% upper confidence interval for pooled standard deviation at baseline for use of full trial sample calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Henry, PH.D., Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ducharme L, Lo C, Hier M, Zeitouni A, Kost K, Mlynarek A, Antoni M, Kuhn E, Owen JE, Heyland D, Platt R, Fuehrmann F, Sadeghi N, Rosberger Z, Frenkiel S, Sultanem K, Shenouda G, Cury F, Henry M. PTSD Coach as an early mobile intervention to improve cancer-related anxiety and psychosocial oncology uptake in patients newly diagnosed with head and neck cancer: pilot randomized controlled trial. Pilot Feasibility Stud. 2024 Dec 21;10(1):153. doi: 10.1186/s40814-024-01556-7. PMID 39709459

DOCUMENTS (1):
  • Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03651570/ICF_000.pdf